CLINICAL TRIAL: NCT02115776
Title: A New Antibiotic Prophylaxis Regimen to Prevent Bacteremia Following Dental Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Pedro DIz DIos, Associate Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PGIDIT05PXIB92501PR
Record Dates: First submitted 2014-04-08; First posted 2014-04-16 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Bacteremia
Keywords: bacteremia; prophylaxis; antibiotics; dentistry
MeSH Terms: conditions — Bacteremia | interventions — Amoxicillin-Potassium Clavulanate Combination; Amoxicillin; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control (No Intervention): Receiving no prophylaxis
- Amoxicillin (Active Comparator): Receiving 2 g Amoxicillin intravenously before any dental manipulation and following endotracheal intubation
  Interventions: Drug: Amoxicillin
- Amoxicillin-Potassium Clavulanate (Experimental): Receiving 1000/200mg Amoxicillin-Potassium Clavulanate i.v. before any dental manipulation and following endotracheal intubation
  Interventions: Drug: Amoxicillin-Potassium Clavulanate
- Chlorhexidine (CHX) (Active Comparator): Receiving a single 0.2% Chlorhexidine (CHX) mouthwash for 30 seconds before any dental manipulation and following endotracheal intubation
  Interventions: Drug: Chlorhexidine
- Amoxicillin-Potassium Clavulanate-CHX (Experimental): Receiving 1000/200mg Amoxicillin-Potassium Clavulanate i.v. and a single 0.2% Chlorhexidine (CHX) mouthwash for 30 seconds before any dental manipulation and following endotracheal intubation
  Interventions: Drug: Amoxicillin-Potassium Clavulanate; Drug: Chlorhexidine

INTERVENTIONS:
Drug: Amoxicillin-Potassium Clavulanate — Administer Amoxicillin-Potassium Clavulanate following endotracheal intubation prior to single tooth-extraction
  Other Names: AMOXICILINA + ACIDO CLAVULANICO SANDOZ EFG (code 600144)
  Arms: Amoxicillin-Potassium Clavulanate; Amoxicillin-Potassium Clavulanate-CHX
Drug: Amoxicillin — Administer Amoxicillin following endotracheal intubation prior to single tooth-extraction
  Other Names: AMOXICILINA SANDOZ EFG (code 694688)
  Arms: Amoxicillin
Drug: Chlorhexidine — Administer Chlorhexidine Digluconate following endotracheal intubation prior to single tooth extraction
  Other Names: Oraldine Perio (code 375725)
  Arms: Amoxicillin-Potassium Clavulanate-CHX; Chlorhexidine (CHX)

SUMMARY:
The aim of this study is to evaluate the efficacy of prophylactic dosage with amoxicillin (AMX), amoxicillin-clavulanate (AMX-CLV), and a combination of amoxicillin-clavulanate and a chlorhexidine mouthwash (AMX-CLV-CHX) in the prevention of bacteremia following dental extractions.

The study hypothesis is that an antimicrobial regimen with amoxicillin-clavulanate will show higher effectiveness in reducing the prevalence and duration of bacteremia following dental extractions, than that achieved with the classical amoxicillin regimen.

DETAILED DESCRIPTION:
PURPOSE: Despite the controversy about the risk of developing bacterial endocarditis of oral origin, numerous Expert Committees in different countries continue to publish prophylactic regimens. To date, the literature is unclear about the role of antimicrobial prophylaxis in the prevention of bacteremia following dental procedures. The aim of this study is to evaluate the efficacy of prophylactic dosage with amoxicillin (AMX), amoxicillin-clavulanate (AMX-CLV), and a combination of amoxicillin-clavulanate and a CHX mouthwash (AMX-CLV-CHX) in the prevention of bacteremia following dental extractions.

SELECTION OF THE STUDY GROUP AND STUDY DESIGN: The study group will comprise patients who, for behavioral reasons (autism, learning disabilities, phobias, etc.), will undergo dental extractions under general anesthesia in the Santiago de Compostela University Hospital (Santiago de Compostela, Spain). The following exclusion criteria will be applied: age under 18 years; body weight under 40 kg; receipt of antibiotics in the previous 3 months; routine use of oral antiseptics; a history of allergy or intolerance to AMX, CHX or AMX-CLV; any type of congenital or acquired immunodeficiency; or any known risk factor for bacterial endocarditis. By applying these criteria, 200 patients will be selected and will be randomly distributed into 5 study groups: control group (receiving no prophylaxis), AMX group (receiving 2 g AMX i.v.), AMX-CLV group (receiving 1000/200mg AMX-CLV i.v.), CHX group (receiving a single 0.2% CHX mouthwash for 30 seconds), and AMX-CLV-CHX group (receiving 1000/200mg AMX-CLV i.v. and a single 0.2% CHX mouthwash for 30 seconds).

COLLECTION OF SAMPLES FOR BLOOD CULTURE: To determine the prevalence of bacteremia, a peripheral venous blood sample (10 ml) will be drawn from each patient at the baseline (before any dental manipulation but after nasotracheal intubation) and 30 s, 15 min, and 1 h after the final dental extraction. Samples will be inoculated in BACTEC plus (Becton Dickinson and Company, Sparks, MD) aerobic and anaerobic blood culture bottles, and will be processed in the Bactec 9240 (Becton Dickinson).

MICROBIOLOGICAL ANALYSIS OF BLOOD CULTURES: A Gram stain will be performed on each positive blood culture. The positive blood cultures in the aerobic media will be subcultured on blood agar and chocolate agar in an atmosphere of 5 to 10% carbon monoxide and on MacConkey agar under aerobic conditions. The same protocol will be used for the positive blood cultures in the anaerobic media, with subculture on Schaedler agar and incubation in an anaerobic atmosphere. The bacteria isolated will be identified by using the battery of biochemical tests provided with the Vitek system for Gram-positive bacteria, Neisseria spp., Haemophilus spp., and obligate anaerobic bacteria. The viridans group streptococci will be classified into five groups, the Streptococcus mitis, S. anginosus, S. salivarius, S. mutans, and S. bovis groups, by applying the Ruoff criteria. Facklam's criteria will be used to identify unusual Streptococcus spp. and other gram-positive cocci in chains.

The subculture and further identification of the isolated bacteria will be performed by conventional microbiological techniques. The collection, handling, and transport of the blood samples for blood culture will be performed according to the recommendations of the Spanish Society of Infectious Diseases and Clinical Microbiology.

.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have at least 10 teeth
* Subjects must have the need for a dental extraction under general anesthesia (for behavioral reasons)
* Subjects will be recruited regardless of the extent and severity of their dental and/or periodontal disease

Exclusion Criteria:

* Age under 18 years
* Body weight under 40 kg
* Receipt of antibiotics in the previous 3 months
* Routine use of oral antiseptics
* A history of allergy or intolerance to amoxicillin
* A history of allergy or intolerance to chlorhexidine
* A history of allergy or intolerance to amoxicillin-clavulanate
* Any type of congenital or acquired immunodeficiency
* Any known risk factor for bacterial endocarditis
* Any known risk factor for prolonged bleeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of participants receiving a prophylactic dosage with amoxicillin-clavulanate i.v. with bacteremia following dental extractions | Changes from baseline in prevalence of bacteremia at 30 seconds, 15 minutes and 1 hour after the final dental extraction
  Percentage of participants receiving a prophylactic dosage with amoxicillin-clavulanate i.v. with bacteremia confirmed by microbiological analysis at 30 seconds, 15 minutes and 1 hour after the final dental extraction

SECONDARY OUTCOMES:
Number of participants receiving a prophylactic dosage with amoxicillin i.v. (following the American Heart Association´s guidelines) with bacteremia after dental extractions | Changes from baseline in prevalence of bacteremia at 30 seconds, 15 minutes and 1 hour after the final dental extraction
  Percentage of participants receiving a prophylactic dosage with amoxicillin i.v. with bacteremia confirmed by microbiological analysis at 30 seconds, 15 minutes and 1 hour after the final dental extraction

OTHER OUTCOMES:
Number of control participants with bacteremia following dental extractions under general anesthesia | Changes from baseline in prevalence of bacteremia at 30 seconds, 15 minutes and 1 hour after the final dental extraction
  Percentage of control participants with bacteremia confirmed by microbiological analysis at 30 seconds, 15 minutes and 1 hour after the final dental extraction

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Diz, MD,DDS,PhD, Study Chair — Universidad de Santiago (Grupo OMEQUI-2117); Hospital Clínico Universitario de Santiago; Jacobo Limeres, DDS,PhD, Study Director — Universidad de Santiago (Grupo OMEQUI-2117); Javier Alvarez, MD,DDS, Principal Investigator — Universidad de Santiago (Grupo OMEQUI-2117); Javier F Feijoo, MD,DDS,PhD, Principal Investigator — Universidad de Santiago (Grupo OMEQUI-2117); Hospital Clínico Universitario de Santiago; Marcio Diniz, DDS,PhD, Principal Investigator — Universidad de Santiago (Grupo OMEQUI-2117); Mercedes Outumuro, DDS,PhD, Principal Investigator — Universidad de Santiago (Grupo OMEQUI-2117); Juan Medina, MD,Anest,PhD, Principal Investigator — Hospital Clínico Universitario de Santiago; Miguel Castro, MD,DDS, PhD, Principal Investigator — Universidad de Santiago (Grupo OMEQUI-2117); Maximiliano Alvarez, MD,Micro,PhD, Principal Investigator — Hospital Clínico Universitario de Vigo
Locations (2):
- Spain (2):
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Santiago de Compostela University Hospital, Santiago de Compostela, Coruña

REFERENCES:
- [Background] Tomas I, Alvarez M, Limeres J, Potel C, Medina J, Diz P. Prevalence, duration and aetiology of bacteraemia following dental extractions. Oral Dis. 2007 Jan;13(1):56-62. doi: 10.1111/j.1601-0825.2006.01247.x. PMID 17241431
- [Background] Tomas I, Pereira F, Llucian R, Poveda R, Diz P, Bagan JV. Prevalence of bacteraemia following third molar surgery. Oral Dis. 2008 Jan;14(1):89-94. doi: 10.1111/j.1601-0825.2006.01359.x. PMID 18173454
- [Background] Valdes C, Tomas I, Alvarez M, Limeres J, Medina J, Diz P. The incidence of bacteraemia associated with tracheal intubation. Anaesthesia. 2008 Jun;63(6):588-92. doi: 10.1111/j.1365-2044.2008.05449.x. PMID 18477269
- [Background] Pineiro A, Tomas I, Blanco J, Alvarez M, Seoane J, Diz P. Bacteraemia following dental implants' placement. Clin Oral Implants Res. 2010 Sep;21(9):913-8. doi: 10.1111/j.1600-0501.2010.01928.x. PMID 20701619
- [Background] Tomas I, Diz P, Tobias A, Scully C, Donos N. Periodontal health status and bacteraemia from daily oral activities: systematic review/meta-analysis. J Clin Periodontol. 2012 Mar;39(3):213-28. doi: 10.1111/j.1600-051X.2011.01784.x. Epub 2011 Sep 15. PMID 22092606
- [Background] Diz Dios P, Tomas Carmona I, Limeres Posse J, Medina Henriquez J, Fernandez Feijoo J, Alvarez Fernandez M. Comparative efficacies of amoxicillin, clindamycin, and moxifloxacin in prevention of bacteremia following dental extractions. Antimicrob Agents Chemother. 2006 Sep;50(9):2996-3002. doi: 10.1128/AAC.01550-05. PMID 16940094
- [Background] Diz Dios P. Infective endocarditis prophylaxis. Oral Dis. 2014 May;20(4):325-8. doi: 10.1111/odi.12221. Epub 2014 Jan 13. PMID 24373017
- [Derived] Limeres Posse J, Alvarez Fernandez M, Fernandez Feijoo J, Medina Henriquez J, Lockhart PB, Chu VH, Diz Dios P. Intravenous amoxicillin/clavulanate for the prevention of bacteraemia following dental procedures: a randomized clinical trial. J Antimicrob Chemother. 2016 Jul;71(7):2022-30. doi: 10.1093/jac/dkw081. Epub 2016 Mar 29. PMID 27029851